CLINICAL TRIAL: NCT05366296
Title: A Randomized, Observer-Blinded, Placebo-Controlled Phase I Study to Evaluate the Safety, Reactogenicity, and Immunogenicity of One Dose Booster by A Lyophilized COVID-19 mRNA Vaccine in Adults Aged 18 to 60 Years
Brief Title: Safety, Reactogenicity, and Immunogenicity Study of a Lyophilized COVID-19 mRNA Vaccine
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: business stragety
Sponsor: Wuhan Recogen Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R520A101; NCT05351450 (obsolete NCT alias)
Record Dates: First submitted 2022-05-03; First posted 2022-05-09 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: COVID-19 Pandemic
MeSH Terms: conditions — COVID-19 | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- : A Lyophilized COVID-19 mRNA Vaccine(RH109) (Active Comparator): Participants received A Lyophilized COVID-19 mRNA Vaccine 0.5ml reconstituted by sterile water, 1 shots at Day0, intramuscular injection
  Interventions: Biological: A Lyophilized COVID-19 mRNA Vaccine
- Placebo control (Placebo Comparator): Participants received placebo of 0.5ml normal saline (0.9% sodium chloride solution), 1 shots at Day0, intramuscular injection
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: A Lyophilized COVID-19 mRNA Vaccine — Active substance: NTD-RBD derived from S protein of Omicron variant Excipient: ALC-0315 (4- hydroxybutyl)azanediyl)bis(hexane-6,1-diyl)bis(2- hexyldecanoate), ALC-0159 (2-[(polyethylene glycol)-2000]-N, N-ditetradecylacetamide), DSPC [1,2- distearoyl-sn-glycero-3-phosphocholine], Cholesterol, Trometamol and Sucrose
  Other Names: RH109
  Arms: : A Lyophilized COVID-19 mRNA Vaccine(RH109)
Biological: Placebo — Normal saline (0.9% sodium chloride solution
  Other Names: Normal saline
  Arms: Placebo control

SUMMARY:
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) is the pathogen that causes a coronavirus-associated acute respiratory disease called coronavirus disease 19 (COVID-19), which is spreading all over the world. This virus can cause acute respiratory distress syndrome (ARDS) with a high fatality rate. In this phase I first-in-human clinical trial, healthy volunteers in two dose cohorts will be vaccinated Lyophilized COVID-19 mRNA Vaccine (RH109) The aim of the study is to assess the safety, reactogenicity and Immunogenicity of the candidate vaccine and to characterize its immunogenicity.

DETAILED DESCRIPTION:
Participants will be enrolled into 2 ascending dose (RH109 low-dose 25 μg, high-dose 50 μg) cohorts randomly. Approximately 24 eligible participants, 12 for each cohort, will be randomized with a 3:1 ratio (RH109 : Placebo). The study will progress in a sequential manner, with the low-dose cohort being enrolled and dosed first. Dose escalation from low-dose to high-dose cohort is contingent on a review of safety data of the low-dose cohort through to 7 days following the vaccination by a Safety Monitoring Committee (SMC)

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 60 years (included) at screening.
2. Have a body mass index (BMI) between 18.5 and 35.0 kg/m2 (included)
3. Able and willing to comply with all study requirements.
4. Willing to allow the Investigator to discuss the volunteers'participant's medical history with his/her general practitioner/personal doctors and access all medical records which are relevant to study procedures.
5. Participants who are of general good health, or with medically stable, well-controlled comorbidities according to the Investigator's assessment, based on medical history at the time of screening and clinical evaluations.
6. Have completed three doses vaccination by any mRNA COVID-19 vaccine 3~12 months (90~365 days, included) prior to the study vaccination.
7. Females of childbearing potential who are involved in heterosexual sexual activity, must be willing to practice continuous effective contraception until 90 days after the study vaccination and have negative pregnancy tests before study vaccination.

   * Nonchildbearing potential is defined as surgically sterile (history of bilateral tubal ligation, bilateral oophorectomy, hysterectomy) or postmenopausal (defined as amenorrhea for ≥ 12 consecutive months prior to Screening without an alternative medical cause). A follicle-stimulating hormone (FSH) level may be measured at the discretion of the Investigator to confirm postmenopausal status.
   * The effective contraceptive methods include sexual abstinence or adequate contraceptive measures such as intrauterine or implanted contraceptive device, oral contraceptives, injected or implanted contraceptives, sustained-release topical contraceptives, condoms (male), diaphragm, and cervical cap, etc.
8. Males participating in this study who are involved in heterosexual sexual activity must agree to practice adequate contraception (as described above) and refrain from donating sperm until 90 days after the study vaccination.
9. Agreement to refrain from blood donation during the study from time of informed consent until end of study visit.
10. Provide written informed consent form (ICF) prior to any study screening activity.

Exclusion Criteria:

1. Laboratory confirmed SARS-CoV-2 infection (history), defined by the result of SARS-CoV-2 RT-PCR assay is positive, and/or SARS-CoV-2 nucleocapsid protein antibody is positive.
2. Documented medical history of COVID-19 disease.
3. Fever (oral temperature ≥ 37.5°C / axillary temperature ≥ 37.3°C) on the day of vaccination. Or having fever within 72 hours before the vaccination.
4. Having abnormal results of clinical laboratory testing during screening, which is judged by the Investigator to be clinically significant, including hematology, clinical chemistry, urinalysis, and coagulation.
5. History of severe allergic disease or reactions likely to be exacerbated by any component of investigational vaccine, such as allergic shock, allergic laryngeal edema, allergic purpura, thrombocytopenic purpura, local hypersensitive necrosis reaction (Arthus reaction), prior history of serious adverse reaction to any vaccine or drug, such as allergy, urticaria eczema, dyspnea, and angioneurotic edema.
6. Having malignant tumor (except for skin basal cell carcinoma or carcinoma uterine cervix in situ), immune disease (e.g., documented human immunodeficiency virus [HIV] infection, systemic lupus erythematosus, rheumatoid arthritis, alienia or splenectomy, and other immune disease that may influence immune response at the Investigator's discretion).
7. Having severe and/or uncontrolled conditions, including but not limited to, acute infectious disease, cardiovascular disease (including history of myocarditis or pericarditis), respiratory disease, gastrointestinal disease, liver disease, renal disease, hematology disease, endocrine disorder, psychiatric condition and neurological illness. Mild/moderate well-controlled comorbidities are allowed to participate.
8. Having bleeding disorder (e.g. factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following intramuscular injections or venipuncture.
9. Received immunosuppressant or other immunomodulators, antiallergic therapy, or cytotoxicity therapy for 14 or more consecutive days within 6 months before the study vaccination. Local administration of immunosuppressant or immunomodulator is allowed (e.g., ointment, eye drops, inhalation, or nasal spray). Drugs for local administration should not be given at a dose over the recommended level in package insert or participants should have no signs of systemic exposure.
10. Administration of immunoglobulin and/or blood product within 3 months before the study vaccination or plan to use that during the study.
11. Continuous use of anticoagulants, such as coumarins and related anticoagulants (e.g., warfarin) or novel oral anticoagulants (e.g., apixaban, rivaroxaban, dabigatran and edoxaban).
12. Used other investigational drug or interventional device within 1 month before the study vaccination or plan to use that during the study, or are using other investigational drug or are within 5 half-lives after the last dose of the investigational drug.
13. Used a subunit or inactivated vaccine within 14 days or an attenuated live vaccine within 1 month (30 days) before the study vaccination, or plan to receive any other vaccines except for the seasonal influenza vaccine, or emergency use authorized vaccines during the study.
14. Prior receipt of any investigational or licensed COVID-19 vaccine except for the mRNA vaccines according to the protocol, or plan to receive any COVID-19 vaccine except for the investigational product (IP)s during the study stage.
15. Suspected or known current alcohol or drug dependency.
16. Having contraindications for intramuscular injection or intravenous blood sampling.
17. Pregnancy, lactation or plan to become pregnant within 90 days after receiving study vaccine.
18. Staff of study site, sponsor, and contract research organization (CRO) taking part in study conduct.
19. At the Investigator's discretion, any other significant disease, disorder or finding that may increase the risk because of participation in the study, or prevent from participation in the study, or impair interpretation of the study data

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
The occurrence of solicited local and systemic adverse events (AEs) within 7 days after the booster vaccination | Within 7days after each does
The occurrence of unsolicited AEs within 28 days after the booster vaccination. | Time Frame: within 28 days after the booster vaccination
The occurrence of serious adverse events (SAEs) and adverse events of special interest (AESIs) until 6 months after the booster vaccination | Until 6 months after the booster vaccination

SECONDARY OUTCOMES:
Geometric mean titer (GMT) of live-virus neutralizing antibody against SARS-CoV-2 Omicron variant (e.g., BA.1 and BA.2) and SARS-CoV-2 prototype | At 14 days, 28 days, 3 months, and 6 months after the booster vaccination.
Seroconversion rate (SCR) of live-virus neutralizing antibody against SARS-CoV-2 Omicron variant (e.g., BA.1 and BA.2) and SARS-CoV-2 prototype | At 14 days, 28 days, 3 months and 6 months after the booster vaccination.
Geometric mean increase (GMI) of live-virus neutralizing antibody against SARS-CoV-2 Omicron variant (e.g., BA.1 and BA.2) and SARS-CoV-2 prototype | At 14 days, 28 days, 3 months, and 6 months after the booster vaccination.
The GMT of anti-N-terminal domain (NTD) and anti-receptor binding domain (RBD) specific IgG at 14 days, 28 days, 3 months and 6 months after the booster vaccination. | At 14 days, 28 days, 3 months and 6 months after the booster vaccination.
The SCR of anti-N-terminal domain (NTD) and anti-receptor binding domain (RBD) specific IgG at 14 days, 28 days, 3 months and 6 months after the booster vaccination. | At 14 days, 28 days, 3 months and 6 months after the booster vaccination.
The GMI of anti-N-terminal domain (NTD) and anti-receptor binding domain (RBD) specific IgG at 14 days, 28 days, 3 months and 6 months after the booster vaccination | At 14 days, 28 days, 3 months and 6 months after the booster vaccination.

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data (IPD) available